CLINICAL TRIAL: NCT06922253
Title: An Open Label, Balanced, Randomized, Single Dose, Two Treatment, Two Sequence, Four Period, Full-replicate, Oral Bioequivalence Study of Sacubitril and Valsartan 97 mg/103 mg Tablets of Ç.O.S.B., Karaağaç Mahallesi Fatih, Bulvarı No:32, Kapaklı/TEKİRDAĞ and Entresto® (Sacubitril and Valsartan) 97 mg/103 mg Tablets of Novartis Europharm Limited, Irija in Healthy, Adult, Human Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study to Compare Sacubitril and Valsartan Tablets (97mg/103mg) Versus Entresto® (Sacubitril and Valsartan) Tablets (97 mg/103 mg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 24-VIN-0563
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — sacubitril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril and Valsartan Tablets (Experimental): Sacubitril and Valsartan 97 mg / 103 mg Tablets
  Interventions: Drug: Sacubitril and Valsartan-Test product
- Entresto® (Sacubitril and Valsartan) Tablets (Experimental): Entresto® (Sacubitril and Valsartan) 97 mg / 103 mg Tablets
  Interventions: Drug: Sacubitril and Valsartan-Reference product

INTERVENTIONS:
Drug: Sacubitril and Valsartan-Test product — 1 tablet of 97 mg Sacubitril / 103 mg Valsartan
  Arms: Sacubitril and Valsartan Tablets
Drug: Sacubitril and Valsartan-Reference product — 1 tablet of 97 mg Sacubitril / 103 mg Valsartan
  Arms: Entresto® (Sacubitril and Valsartan) Tablets

SUMMARY:
An open label, balanced, randomized, single dose, two treatment, two sequence, four period, full-replicate, oral bioequivalence Study of Sacubitril and Valsartan 97 mg/103 mg Tablets of HUMANİS SAĞLIK ANONİM ŞİRKETİ Ç.O.S.B., Karaağaç Mahallesi Fatih, Bulvarı No:32, Kapaklı/TEKİRDAĞ and Entresto® (Sacubitril and Valsartan) 97 mg/103 mg Tablets of Novartis Europharm Limited, Irija in healthy, adult, human subjects under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 45 years (both inclusive).
* Subjects' weight within normal range according to normal values for Body Mass Index (between 18.50 and 30.00 kg/m2) (both inclusive) with minimum of 45 kg weight.
* Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within the clinically acceptable range.
* Subject with Creatinine Clearance ≥80 ml/min.
* Subjects having clinically acceptable 12-lead electrocardiogram (ECG).
* Subjects having clinically acceptable chest X-Ray (PA view), if taken.
* Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
* Subjects having negative urine alcohol test / breath alcohol test.
* Non-smokers.
* Subjects willing to adhere to the protocol requirements and to provide written informed consent.
* For male Subjects:

Subjects willing to follow approved birth control methods (a double barrier method) for the duration of the study as judged by the investigator(s), such as (a double barrier method) condom with spermicide, Condom with diaphragm, or abstinence. Subjects willing to refrain from donating sperm during the study period

- For Female Subjects: Female of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as intrauterine device (IUD), abstinence, bilateral tubal ligation or double barrier contraception, i.e., condom + diaphragm, condom + spermicidal or foam Postmenopausal for at least 1 year, or if less than 1 year, then following acceptable contraceptive measures as mentioned above

* Subjects having negative urine pregnancy test at screening and negative serum β-hCG pregnancy test on admission day of period 01 (only for female subjects).
* Female Subjects who are non-pregnant and non-lactating.

Exclusion Criteria:

* Subjects having hypersensitivity to Sacubitril and Valsartan or related class of drugs or any of its excipients or heparin.
* Subject with the serum potassium level >5.4 mmol/l during screening.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, urogenital or psychiatric disease or disorder.
* Subjects who undergone any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 30 days prior to admission in period 01.
* History or presence of alcoholism or drug abuse.
* History or presence of asthma, urticaria or other significant allergic reactions.
* History or presence of significant gastric and/or duodenal ulceration.
* History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
* History or presence of cancer or basal or squamous cell carcinoma.
* Subject having difficulty with donating blood.
* Subjects having difficulty in swallowing solid dosage form like tablets or capsules.
* Use of any prescribed medication or OTC medication including vaccines, vitamins and herbal remedies during last 30 days prior to admission in period 01.
* Subject having major illness within past 03 months.
* Volunteer who have donated blood (1 unit) or participation in a drug research study within past 90 days prior to the first dose of the study drug.
* Consumption of xanthine-containing products, tobacco containing products or alcohol or any alcohol containing products within 48.00 hours prior to admission in period 01.
* Consumption of grapefruit or grapefruit juice containing products within 72.00 hours prior to admission of period 01.
* Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
* History or presence of significant easy bruising or bleeding.
* History or presence of significant recent trauma.
* Subjects who have been on an abnormal diet (for whatever reason) during the four weeks preceding the study.
* Female subjects who are currently breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 48.00 hours
  If the intra-subject CV of the reference formulation for Cmax is less than or equal to 30%, the conventional acceptance range of 80.00% - 125.00% for bioequivalence will be applied to Cmax.
Area Under the Curve from time zero to time of last measurable concentration (AUC0-t) | 48.00 hours
  For, AUC0-t, acceptance range for bioequivalence is 80.00 - 125.00% for 90% confidence intervals of the geometric least square means ratio (T/R).

SECONDARY OUTCOMES:
Area Under the Curve from time zero to time infinite (AUC0-∞) | 48.00 hours
  descriptive statistics
Time to reach peak plasma concentration (Tmax) | 48.00 hours
  descriptive statistics
Plasma Elimination Half-Life (t1/2) | 48.00 hours
  descriptive statistics
The elimination rate constant (Kel) | 48.00 hours
  descriptive statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Veeda Clinical Research Ltd., Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No